CLINICAL TRIAL: NCT00688649
Title: An Investigation of the Effects of Different Modes of Delivery of Oral Nutritional Supplements in Participants at Risk of Malnutrition - A Pilot Study
Brief Title: Nutritional Supplement Compliance Study
Acronym: NSCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Dr Gary Hubbard, Senior Clinical Research Advisor, Nutricia UK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC200
Record Dates: First submitted 2008-05-27; First posted 2008-06-03 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard ONS
  Interventions: Dietary Supplement: Standard Oral Nutritional Supplement (ONS)
- 2 (Active Comparator): High Energy ONS
  Interventions: Dietary Supplement: High energy Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Dietary Supplement: Standard Oral Nutritional Supplement (ONS) — Standard energy, oral nutritional supplement (a milk style nutritional supplement (1.5kcal/ml, 200ml) containing protein, fat, carbohydrate and micronutrients)
  Arms: 1
Dietary Supplement: High energy Oral Nutritional Supplement (ONS) — High Energy nutritional supplement (a milk style nutritional supplement (2.4kcal/ml, 125ml) containing protein, fat, carbohydrate and micronutrients)
  Arms: 2

SUMMARY:
Disease-related malnutrition is common across healthcare settings in the UK and if left untreated, may have severe consequences. One of the strategies commonly used to combat malnutrition is the use of oral nutritional supplements (ONS). However, there is uncertainty about the optimal way of delivering ONS to patients to maximize compliance and nutrient intake.

This randomised study will investigate the effect of different modes of delivery (ad libitum versus instructions on timing/serving volume) of ONS used in addition to the diet on total nutrient intake, compliance, nutritional status and outcome in participants at risk of malnutrition.

Participants will be randomised to receive one of two ONS (high energy or standard) for 4 weeks in addition to food, either taken 'Ad libitum', or according to instruction on what to take and when. The primary outcome measure is nutrient intake. Secondary outcome measures include compliance and acceptability of ONS, appetite, anthropometry, muscle strength, quality of life and gastro-intestinal tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 18 years
* At risk of malnutrition (medium or high risk of malnutrition with 'Malnutrition Universal Screening Tool', 'MUST' score ≥ 1)
* Competent to provide written informed consent and able to answer questions
* No requirement for tube or parenteral feeding
* Willingness to take part in the study and to follow the study protocol

Exclusion Criteria:

* Requirement for tube or parenteral nutrition
* Participants receiving palliative care
* Participants with chronic renal disease requiring dialysis
* Participants with liver failure
* Participants that are pregnant or lactating
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Nutrient intake (energy, protein and micronutrients) | 4 weeks

SECONDARY OUTCOMES:
Compliance with ONS | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Fumi, Study Director — Nutricia UK
Locations (1):
- Royal United Hospital, Nutrition and Dietetics Dept, Bath, Wiltshire, United Kingdom